CLINICAL TRIAL: NCT00742430
Title: Assessment of Aspirin and Clopidogrel Resistance in Ischemic Heart Disease Using Multiplate Function Analyser and it's Correlation With Major Adverse Cardiac Events
Brief Title: Resistance on Antithrombotic Drugs in Ischemic Heart Disease
Status: Completed | Type: Observational
Sponsor: University of Zagreb (Other)
Responsible Party: Principal Investigator, Davor Milicic, prof. dr. sc. F.E.S.C., University of Zagreb
Other Study IDs: 108-1081875-1993
Record Dates: First submitted 2008-08-26; First posted 2008-08-27 (Estimated); Last update posted 2012-02-14 (Estimated); Status verified 2012-02

CONDITIONS: Coronary Artery Disease
Keywords: aspirin resistance; coronary artery disease; clopidogrel resistance; major adverse cardiac events; multiplate platelet function analyser; percutaneous coronary intervention
MeSH Terms: conditions — Coronary Artery Disease; Cardiovascular Diseases | interventions — Stents

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Resistant: patients who are resistant to standard antithrombotic drugs
  Interventions: Procedure: PCI
- Nonresistant: patients who are not resistant to standard dual antithrombotic drugs
  Interventions: Procedure: PCI

INTERVENTIONS:
Procedure: PCI — percutaneous coronary intervention in stable coronary artery disease
  Other Names: stenting; PTCA; balloon dilatation

SUMMARY:
The purpose of this study is to determine whether aspirin and clopidogrel resistance measured with Multiplate function analyser has a good correlation with incidence of major adverse cardiac events in patients with coronary artery disease (CAD).

DETAILED DESCRIPTION:
Our plan is to enroll 180 patients with diagnosed CAD who electively undergo percutaneous coronary intervention (PCI). Blood samples will be taken just before the procedure and one day after the procedure and analysed on Multiplate function analyser. Assessing aspirin and clopidogrel resistance incidence using Multiplate platelet function analyzer we will also try to find resistance correlation with the incidence of major adverse cardiac events in a one year follow up.

ELIGIBILITY:
Inclusion Criteria:

* Elective PCI
* > 7 days on aspirin 100mg therapy before the intervention
* > 7 days on clopidogrel 75mg therapy before the intervention

Exclusion Criteria:

* Loading dose of clopidogrel
* < 7 days on aspirin therapy before the intervention
* Myocardial infarction less than 30 days before the intervention
* Cerebrovascular incident less that three months before the intervention
* Haemorrhagic diathesis
* Trc < 100
* Htc < 30%
* Creatinine > 140

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: patients with coronary artery disease
Sampling Method: Non-Probability Sample
Enrollment: 141 (Actual)
Dates: Start 2009-02; Study Completion 2011-08 (Actual)

PRIMARY OUTCOMES:
Major adverse coronary event | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Davor Milicic, prof.dr.sc., Principal Investigator — Clinic of Cardiovascular Diseases, Clinical Medical Centre Rebro, Zagreb, Croatia; Bosko Skoric, dr., Study Chair — Clinic of Cardiovascular Diseases, Clinical Medical Centre Rebro, Zagreb, Croatia
Locations (1):
- Clinic of Cardiovascular Diseases, Clinical Medical Centre Rebro, Zagreb, Croatia